CLINICAL TRIAL: NCT05222802
Title: A Phase 1 Study to Evaluate the CNS-Penetrant EGFR/ERBB1 Inhibitor ERAS-801 in Patients With Recurrent Glioblastoma (THUNDERBBOLT-1)
Brief Title: A Study to Evaluate ERAS-801 in Patients With Recurrent Glioblastoma (THUNDERBBOLT-1)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Katmai Pharmaceuticals Inc. (Industry)
Collaborators: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-801-01
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; EGFR; epidermal growth factor receptor; alteration; ERBB1
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation (Part 1) (Experimental): ERAS-801 will be orally administered to study participants with recurrent GBM in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-801
- Dose Expansion (Part 2) (Experimental): ERAS-801 will be orally administered at the recommended dose (as determined from Part 1) to study participants with recurrent GBM harboring alterations in EGFR.
  Interventions: Drug: ERAS-801

INTERVENTIONS:
Drug: ERAS-801 — Administered orally

SUMMARY:
* To evaluate the safety and tolerability of escalating doses of ERAS-801 in study participants with recurrent glioblastoma multiforme (GBM).
* To determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) of ERAS-801.
* To evaluate the antitumor activity of ERAS-801.
* To evaluate the PK profile of ERAS-801.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter clinical study evaluating ERAS-801 as a monotherapy. The study will initially commence with dose escalation of ERAS-801 in study participants with recurrent GBM. Once the MTD and/or RD has been determined from dose escalation, then dose expansion of ERAS-801 may commence in study participants with recurrent GBM harboring alterations in epidermal growth factor receptor (EGFR).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing and able to give written informed consent
* Diagnosis of Glioblastoma, IDH WT as defined by the WHO 2021 criteria
* Adequate organ function
* Willing to comply with all protocol-required visits, assessments, and procedures
* Able to swallow oral medication

Exclusion Criteria:

* Prior treatment with an EGFR inhibitor for Glioblastoma
* Currently enrolled in another therapeutic study
* History of clinically significant cardiovascular disease
* Gastrointestinal conditions that may affect administration/absorption of oral medications
* Have an active infection (bacterial, fungal, or viral) requiring systemic therapy
* Pregnant or breastfeeding women
* Any serious underlying medical or psychiatric condition or evidence of any other significant clinical disorder or laboratory finding that renders the patient inappropriate to participate in the study
* Known allergies, hypersensitivity, or intolerance to ERAS-801 or its excipients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Maximum Tolerated Dose (MTD) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Recommended Dose (RD) | Study Day 1 up to Day 29
  Based on adverse events observed during dose escalation
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs

SECONDARY OUTCOMES:
Plasma concentration (Cmax) | Study Day 1 up to Day 29
  Maximum plasma or serum concentration of ERAS-801
Time to achieve Cmax (Tmax) | Study Day 1 up to Day 29
  Time to achieve maximum plasma or serum concentration of ERAS-801
Area under the curve | Study Day 1 up to Day 29
  Area under the plasma concentration-time curve of ERAS-801
Half-life | Study Day 1 up to Day 29
  Half-life of ERAS-801
Objective Response Rate (ORR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per modified RANO response assessment
Duration of Response (DOR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per modified RANO response assessment
Time to Response (TTR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per modified RANO response assessment

CONTACTS AND LOCATIONS:
Overall Officials: Les Brail, Study Director — Medical Director
Locations (8):
- United States (8):
  - University of California, Los Angeles, Los Angeles, California
  - Miami Cancer Institute-Baptist Heath South Florida, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Sarah Cannon Research Institute (Tennessee Oncology), Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No